CLINICAL TRIAL: NCT00525395
Title: Continuative vs Sequential Phototherapy in Non-segmental Vitiligo Patients
Brief Title: Virus Early Transcription Factor (VETF) Multicenter Phototherapy Protocol
Acronym: VETF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituti Fisioterapici Ospitalieri (Other)
Responsible Party: Dott. Mauro Picardo, Istituto San Gallicano - Roma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VETF01
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-06

CONDITIONS: Vitiligo
Keywords: Phototherapy; Vitiligo scoring system
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Group A: 2 months treatment-1 month no treatment-2 months treatment-1 month no treatment
  Interventions: Genetic: Sequential phototherapy
- B (Active Comparator): Group B: 6 months non-stop treatment.
  Interventions: Procedure: Continuous phototherapy

INTERVENTIONS:
Genetic: Sequential phototherapy — Group A: 2 months treatment-1 month no treatment-2 months treatment-1 month no treatment
  Arms: A
Procedure: Continuous phototherapy — Group B: 6 months non-stop treatment.
  Arms: B

SUMMARY:
Background

Phototherapy UVB TL01 currently represents the first choice in treatment to induce the repigmentation of vitiligo spots. The problem though is that there are no systems or scales which enable an objective evaluation of the therapy, commonly known as percentage of repigmentation.

Recently, a European Task Force (VETF, Vitiligo European Task Force) of experts on vitiligo, within the European Society of Pigmentation, has proposed a gravity classification on the basis of three parameters/standards - extension, progression and the level of depigmentation - and used to classify patients in ten European centres. The aim of the trial is to validate the VETF scoring system set up in relation with the therapeutic answer to the standard treatment for vitiligo and phototherapy.

Leaving aside short term side effects, such as sunrush/erythema and sunburn, which are reversible and infrequent, the main problem with phototherapy is represented by the cumulative long term effects of ultraviolet rays. These can cause premature ageing of the skin (photoaging) and the appearance of skin cancer/neoplasia. Therefore the aim is to get the best results from phototherapy whilst limiting its length.

Aims of the trial:

1. To validate the VETF scoring system. As phototherapy is currently the only universally accepted treatment for vitiligo, it seems logical to test the VETF scoring system first to evaluate the effectiveness of phototherapy.
2. Secondly, the target of this multicentric trial is to compare the effectiveness of two different phototherapy protocols; a first protocol foresees non-stop treatment for 6 months; a second protocol foresees periods of interruption during the treatment. This will help to verify whether interrupting a cycle of phototherapy is useful or not.

This interruption might make the ultraviolet rays more effective 'stimulus on the melanocytes', and may also reduce long term damage caused by phototherapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years old

Exclusion Criteria:

* Phototype I
* Previous treatment with any kind of phototherapy in the last 6 months.
* Patients with counter indications for PUVA or phototherapy (history of skin cancer, pregnancy, etc.).
* Acral vitiligo (only hands and feet are affected).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The percentage of repigmentation on the target lesions will be evaluated at the end of each treatment in both groups. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Picardo, MD, Study Chair — Istituto San Gallicano - Rome - Italy
Locations (1):
- Istituto San Gallicano -, Rome, Rome, Italy